CLINICAL TRIAL: NCT03064074
Title: Multicenter Study to Evaluate Safety of Fresolimumab in Adults With Moderate-to-severe Osteogenesis Imperfecta
Brief Title: Safety of Fresolimumab in the Treatment of Osteogenesis Imperfecta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brendan Lee, Chairman/Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H37912
Record Dates: First submitted 2016-10-13; First posted 2017-02-24 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stage 1 Low dose (Experimental): There are a total of 6 study visits within approximately a 6 month timespan. Investigators will evaluate the safety of a single administration of fresolimumab in adult patients with OI. Subjects will receive a single-dose of 1 mg/kg of fresolimumab (n=4).
  At each study visit, the participant may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  Interventions: Drug: Fresolimumab
- Stage 2 High dose (Experimental): There are a total of 6 study visits within approximately a 6 month timespan. Investigators will evaluate the safety of a single administration of fresolimumab in adult patients with OI. Subjects will receive a single-dose of 4 mg/kg of fresolimumab (n=4).
  At each study visit, the participant may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  Interventions: Drug: Fresolimumab
- Stage 2 Repeat dose every 6 months (Experimental): Fresolimumab will be administered every six months for a total treatment period of 12 months (Total Anticipated n=4). The dose to be administered (1 or 4 mg/kg) will be chosen after completion of Stage 1. The primary Stage 2 endpoint will be safety measures assessed over 12 months. The secondary endpoints will be changes in markers of bone remodeling, bone mineral density, estimated strength.
  At each study visit, participants may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  * Skeletal survey
  * Peripheral quantitative CT (pQCT) of the forearm
  * Quality of Life Surveys
  * Pulmonary function test
  * Walk test
  Interventions: Drug: Fresolimumab
- Stage 2 Repeat doses every 3 months (Experimental): Fresolimumab will be administered every three months for a total treatment period of 12 months (Total anticipated n=4). The dose to be administered (1 or 4 mg/kg) will be chosen after completion of Stage 1. The primary Stage 2 endpoint will be safety measures assessed over 12 months. The secondary endpoints will be changes in markers of bone remodeling, bone mineral density, estimated strength.
  At each study visit, participants may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  * Skeletal survey
  * Peripheral quantitative CT (pQCT) of the forearm
  * Quality of Life Surveys
  * Pulmonary function test
  * Walk test
  Interventions: Drug: Fresolimumab

INTERVENTIONS:
Drug: Fresolimumab — The purpose of this study is to determine if fresolimumab is safe as a treatment for OI. We will evaluate the safety of a single dose of fresolimumab in the 1st stage of the study. We will evaluate the safety of multiple doses of fresolimumab in the 2nd stage of the study. The Investigators will evaluate the effect of the two doses of fresolimumab in Stage 1 on markers of bone turnover and determine the dose that shows the greatest reduction in bone turnover markers compared to no treatment. This dose will be chosen for the repeat dose studies. If there were no significant changes between the bone turnover markers with either dose, the 4 mg/kg dose will be chosen for the repeat dose study.

SUMMARY:
Osteogenesis Imperfecta (OI) is a rare disorder that causes bones to break easily. People with OI may have broken bones with little or no trauma, dentinogenesis imperfecta (DI), and, in adult years, hearing loss. OI can range from very severe to very mild. The current standard-of-care for severe types of OI involves the use of IV medications (bisphosphonates) and surgery to put rods in bones to strengthen them. These therapies, although often life-saving, are new and very little is known about their long-term effects on bone and other body systems.

Transforming growth factor beta (TGF-β) is a protein important in bone formation. Fresolimumab is an antibody that can silence TGF-β . In studies with mice with OI, it has been shown that silencing TGF-β can lead to higher bone mass, quality and strength. The purpose of this study is to determine if fresolimumab is safe in the treatment of OI.

DETAILED DESCRIPTION:
Osteogenesis Imperfecta (OI) is a rare disorder that causes bones to break easily. People with OI may have broken bones with little or no trauma, dentinogenesis imperfecta (DI), and, in adult years, hearing loss. It is seen in both genders and all races. OI can range from very severe to very mild. Individuals with the most severe type of OI may die at birth. People with severe OI who survive may have bowed arms and legs, very short stature and be unable to walk. People with the mildest form of OI may only break bones occasionally and have normal height and lifespan. Breaks can occur in any bone, but are most common in the arms and legs. The current standard-of-care for severe types of OI involves the use of IV medications (bisphosphonates) and surgery to put rods in bones to strengthen them. These therapies, although often life-saving, are new and very little is known about their long-term effects on bone and other body systems.

TGF-β is a protein important in bone formation. Studies have shown that increased TGF-β activity leads to lower bone mass and strength and increased fractures. Fresolimumab is an antibody that can silence TGF-β . In studies with mice with OI, it has been shown that silencing TGF-β can lead to higher bone mass, quality and strength.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed informed consent.
2. Are 18 years or older
3. Have a diagnosis of moderate-to-severe OI based on various clinical features
4. Have genetic mutations that include glycine substitution in COL1A1 or COL1A2, or pathogenic variants in CRTAP, PPIB, or LEPRE1 (if genetic information is unavailable at screening, this may be assessed at screening visit on a clinical or research basis).
5. Females of child-bearing potential must have a negative urine pregnancy test, agree to and have the ability to use acceptable birth control method for entire duration of the study.
6. For Males enrolled in the study, partners must agree to use an acceptable form of birth control for the entire duration of the study.

Exclusion Criteria:

1. Fracture less than 3 months prior to the screening visit.
2. Rodding or instruments that prevents reliable bone mineral density (BMD) assessment.
3. Have a known unhealed fracture involving a long bone.
4. Do not meet laboratory safety requirements such as: Vitamin D < 15 ng/dL Serum albumin-corrected calcium levels below 8 mg/dL, Hemoglobin < 10 g/dL, Platelet count < 75,000mm3;, Prothrombin time/(PT/INR) international normalized ratio > 1.5 times Upper Limit of Normal (ULN), Clinical or laboratory abnormality of Grade III or higher as assessed by CTCAE v4.0 which in the view of investigator would compromise safety.
5. Have an EKG with QTc of > 450 ms
6. Have a known allergy to fresolimumab.
7. Have current clinically significant infection.
8. Have a personal history of basal cell carcinoma, squamous cell carcinoma or keratoacanthomas, a personal history of cancer, recent or remote.
9. Have evidence of untreated cavities or planned invasive dental work during the study period.
10. Have had organ transplantation.
11. Have known or suspected valvular heart disease.
12. Plan to have skeletal surgery in the study period.
13. Have had osteotomy 5 months prior to the screening visit.
14. Being treated with zoledronic acid or pamidronate less than 12 months of screening OR oral bisphosphonates less than 6 months of screening OR teriparatide less than one year of screening.
15. Being treated with systemic glucocorticoids
16. Have autoimmune diseases being treated with glucocorticoids or other biologic agents.
17. Enrolled in another clinical trial and receiving treatment with another investigational agent
18. Pregnant or planning to get pregnant during the study period.
19. Nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh Nagamani, M.D., Study Chair — Baylor College of Medicine; VReid Sutton, M.D., Study Chair — Baylor College of Medicine; Brendan Lee, M.D., Ph.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Oregon Health Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Song IW, Nagamani SC, Nguyen D, Grafe I, Sutton VR, Gannon FH, Munivez E, Jiang MM, Tran A, Wallace M, Esposito P, Musaad S, Strudthoff E, McGuire S, Thornton M, Shenava V, Rosenfeld S, Huang S, Shypailo R, Orwoll E, Lee B. Targeting TGF-beta for treatment of osteogenesis imperfecta. J Clin Invest. 2022 Apr 1;132(7):e152571. doi: 10.1172/JCI152571. PMID 35113812

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Low Dose: There are a total of 6 study visits within approximately a 6 month timespan. Investigators will evaluate the safety of a single administration of fresolimumab in adult patients with OI. Subjects will receive a single-dose of 1 mg/kg of fresolimumab (n=4).
  At each study visit, the participant may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  Fresolimumab: The purpose of this study is to determine if fresolimumab is safe as a treatment for OI. We will evaluate the safety of a single dose of fresolimumab in the 1st stage of the study. We will evaluate the safety of multiple doses of fresolimumab in the 2nd stage of the study. The Investigators will evaluate the effect of the two doses of fresolimumab in Stage 1 on markers of bone turnover and determine the dose that shows the greatest reduction in bone turnover markers compared to no treatment. This dose will be chosen for the repeat dose studies. If there were no significant changes between the bone turnover markers with either dose, the 4 mg/kg dose will be chosen for the repeat dose study.
- Stage 2 High Dose: There are a total of 6 study visits within approximately a 6 month timespan. Investigators will evaluate the safety of a single administration of fresolimumab in adult patients with OI. Subjects will receive a single-dose of 4 mg/kg of fresolimumab (n=4).
  At each study visit, the participant may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  Fresolimumab: The purpose of this study is to determine if fresolimumab is safe as a treatment for OI. We will evaluate the safety of a single dose of fresolimumab in the 1st stage of the study. We will evaluate the safety of multiple doses of fresolimumab in the 2nd stage of the study. The Investigators will evaluate the effect of the two doses of fresolimumab in Stage 1 on markers of bone turnover and determine the dose that shows the greatest reduction in bone turnover markers compared to no treatment. This dose will be chosen for the repeat dose studies. If there were no significant changes between the bone turnover markers with either dose, the 4 mg/kg dose will be chosen for the repeat dose study.
- Stage 2 Repeat Dose Every 6 Months: Fresolimumab will be administered every six months for a total treatment period of 12 months (n=4). The dose to be administered (1 or 4 mg/kg) will be chosen after completion of Stage 1. The primary Stage 2 endpoint will be safety measures assessed over 12 months. The secondary endpoints will be changes in markers of bone remodeling, bone mineral density, estimated strength.
  At each study visit, participants may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  * Skeletal survey
  * Peripheral quantitative CT (pQCT) of the forearm
  * Quality of Life Surveys
  * Pulmonary function test
  * Walk test
  Fresolimumab: The purpose of this study is to determine if fresolimumab is safe as a treatment for OI. We will evaluate the safety of a single dose of fresolimumab in the 1st stage of the study. We will evaluate the safety of multiple doses of fresolimumab in the 2nd stage of the study. The Investigators will evaluate the effect of the two doses of fresolimumab in Stage 1 on markers of bone turnover and determine the dose that shows the greatest reduction in bone turnover markers compared to no treatment. This dose will be chosen for the repeat dose studies. If there were no significant changes between the bone turnover markers with either dose, the 4 mg/kg dose will be chosen for the repeat dose study.
- Stage 2 Repeat Doses Every 3 Months: Fresolimumab will be administered every three months for a total treatment period of 12 months (n=4). The dose to be administered (1 or 4 mg/kg) will be chosen after completion of Stage 1. The primary Stage 2 endpoint will be safety measures assessed over 12 months. The secondary endpoints will be changes in markers of bone remodeling, bone mineral density, estimated strength.
  At each study visit, participants may have the following testing done:
  * Physical exam
  * Vitals
  * Blood draw for safety labs, pharmacokinetics, etc
  * If the participant is female, she will have a pregnancy test
  * EKG
  * DXA
  * Infusion of the study drug
  * Skeletal survey
  * Peripheral quantitative CT (pQCT) of the forearm
  * Quality of Life Surveys
  * Pulmonary function test
  * Walk test
  Fresolimumab: The purpose of this study is to determine if fresolimumab is safe as a treatment for OI. We will evaluate the safety of a single dose of fresolimumab in the 1st stage of the study. We will evaluate the safety of multiple doses of fresolimumab in the 2nd stage of the study. The Investigators will evaluate the effect of the two doses of fresolimumab in Stage 1 on markers of bone turnover and determine the dose that shows the greatest reduction in bone turnover markers compared to no treatment. This dose will be chosen for the repeat dose studies. If there were no significant changes between the bone turnover markers with either dose, the 4 mg/kg dose will be chosen for the repeat dose study.
Period: Overall Study
Arm/Group | Stage 1 Low Dose | Stage 2 High Dose | Stage 2 Repeat Dose Every 6 Months | Stage 2 Repeat Doses Every 3 Months
Started | 4 | 4 | 2 | 1
Completed | 4 | 4 | 2 | 0
Not Completed | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Low Dose | Stage 2 High Dose | Stage 2 Repeat Dose Every 6 Months | Stage 2 Repeat Doses Every 3 Months | Total
Number analyzed (Participants) | 4 | 4 | 2 | 1 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 2 | 1 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 7
  Male | 2 | 1 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 2 | 1 | 8
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 2 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety of single and repeat doses of fresolimumab will be assessed in adult patients with moderate to severe osteogenesis imperfecta
Time Frame: 6 months for single dose study and 12 months for repeat dose study
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Low Dose | Stage 2 High Dose | Stage 2 Repeat Dose Every 6 Months | Stage 2 Repeat Doses Every 3 Months
Number analyzed (Participants) | 4 | 4 | 2 | 1
Participants | 2 | 4 | 2 | 1

2. Secondary Outcome: Percentage Change in Bone Turnover Markers or P1NP, Osteocalcin or Ocn, and C-terminal Telopeptide or CTX
Description: Percentage change in bone turnover markers from baseline to Day 180
Time Frame: 6 months in single dose study and 12 months in repeat dose study
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Stage 1 Low Dose | Stage 2 High Dose | Stage 2 Repeat Dose Every 6 Months | Stage 2 Repeat Doses Every 3 Months
Number analyzed (Participants) | 4 | 4 | 2 | 1
Percent change
  Percentage Change in P1NP | 28.31 (17.44) | 24.95 (17.44) | 118.63 (45.40) | NA (NA) — Only one participant was enrolled. This participant had to be withdrawn due to fracture because of OI and could not complete the study procedures. Thus, the percentage change of P1NP could not be calculated.
  Percentage Change in CTX | 49.89 (29.29) | -4.02 (33.82) | 51.83 (34.56) | NA (NA) — Only one participant was enrolled. This participant had to be withdrawn due to fracture because of OI and could not complete the study procedures. Thus, the percentage change of CTX could not be calculated.
  Percentage change in Osteocalcin | 76.4 (39.1) | -18.6 (39.13) | 83.9 (17.56) | NA (NA) — Only one participant was enrolled. This participant had to be withdrawn due to fracture because of OI and could not complete the study procedures. Thus, the percentage change in Ocn could not be calculated.

ADVERSE EVENTS:
Time Frame: 6 Months for single dose study and 1 year for the multi dose study
Arm/Group | Stage 1 Low Dose | Stage 2 High Dose | Stage 2 Repeat Dose Every 6 Months | Stage 2 Repeat Doses Every 3 Months
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Low Dose (N=4) | Stage 2 High Dose (N=4) | Stage 2 Repeat Dose Every 6 Months (N=2) | Stage 2 Repeat Doses Every 3 Months (N=1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Low Dose (N=4) | Stage 2 High Dose (N=4) | Stage 2 Repeat Dose Every 6 Months (N=2) | Stage 2 Repeat Doses Every 3 Months (N=1)
General Adverse events (Investigations) | 4 (38) | 4 (24) | 2 (13) | 1 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03064074/Prot_SAP_000.pdf